CLINICAL TRIAL: NCT02971371
Title: The Role of Mirror Neuron System in Improving Motor Performance by Using Virtual Reality, as Revealed by EEG: a Randomized Clinical Trial
Brief Title: The Role of MNS in Improving Motor Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Principal Investigator, Rocco Salvatore Calabrò, Principal investigator, IRCCS Centro Neurolesi Bonino Pulejo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 43/2013
Record Dates: First submitted 2016-11-07; First posted 2016-11-22 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Virtual Reality (Experimental): This group performed 40 45-min Lokomat sessions, five times a week, by using a visual feedback showing a Virtual Reality run game where the patient had to collect or avoid objects, to motivate him/her to walk actively.
  Interventions: Device: Lokomat
- Only RAGT (Active Comparator): This groups performed 40 Lokomat sessions (40-45min), five times a week, between 9am and 11am, in this case was not provided an avatar, and a smile indicating the goodness of each leg movement.
  Interventions: Device: Lokomat

INTERVENTIONS:
Device: Lokomat — Both the groups performed 40 45min Lokomat sessions, five times a week, between 9am and 11am. The "RAGT"and "VR" group received a visual feedback showing a VR run game where the patient had to collect or avoid objects, to motivate him/her to walk actively. Each avatar's leg movement corresponded to that performed by the patient. On the other hand, the "RAGT" without "VR" group was not provided an avatar, and a smile indicating the goodness of each leg movement. The biofeedback of the Lokomat gait orthosis is based on the interaction torques between the participant and the orthosis

SUMMARY:
Many studies have demonstrated the usefulness of repetitive task practice by using robotic devices, including Lokomat, for the treatment of lower limb paresis. Virtual reality (VR) has proved to be a valuable tool to improve neurorehabilitation training. Our pilot randomized clinical trial aimed at evaluating the correlation between the modifications of brain oscillations during a VR neurorehabilitative training of gait and the motor function recovery in patients with chronic stroke.

Twenty-four patients suffering from a first unilateral ischemic stroke in the chronic phase were randomized into two groups. One group performed 40 sessions of Lokomat with VR (RAGT+VR) whereas the other group underwent Lokomat without VR (RAGT-VR). Outcomes (clinical, kinematic, and event-related synchronization, ERS, and desynchronization, ERD, at the EEG) were measured before and after the robotic intervention.

The robotic-based rehabilitation combined with VR could be associated with improvements in several measurements of lower limb function, gait, and balance in patient with chronic hemiparesis. Moreover, ERS/ERD analysis can be proposed as a tool to monitor motor performance and to develop non-invasive brain-computer interfaces controlling robotic devices.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥55 years
* A first-ever ischemic supra-tentorial stroke (confirmed by MRI scan) at least 6 months before their enrollment;
* An unilateral hemiparesis, with a Muscle Research Council -MCR- score ≤3
* Ability to follow verbal instructions, with a Mini-Mental State Examination (MMSE) >24
* A mild to moderate spasticity according to a Modified Ashworth Scale (MAS) ≤2
* No severe bone or joint disease
* No history of concomitant neurodegenerative diseases or brain surgery.

Exclusion Criteria:

* Severe cognitive and behavioral impairments
* Severe osteoporosis and previous bone fractures

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-10; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
gait evaluated by Rivermead Mobility Index (RMI) | Six months

SECONDARY OUTCOMES:
Spasticity evaluated by Modified Ashworth Scale (MAS) | Six months

REFERENCES:
- [Derived] Calabro RS, Naro A, Russo M, Leo A, De Luca R, Balletta T, Buda A, La Rosa G, Bramanti A, Bramanti P. The role of virtual reality in improving motor performance as revealed by EEG: a randomized clinical trial. J Neuroeng Rehabil. 2017 Jun 7;14(1):53. doi: 10.1186/s12984-017-0268-4. PMID 28592282